CLINICAL TRIAL: NCT07089875
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of Dotinurad Compared With Allopurinol in Adult Participants With Hyperuricemia Associated With Gout
Brief Title: A Study of Dotinurad Versus Allopurinol in Participants With Gout
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Crystalys Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FYU-981-CRYS-301; 2024-520206-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-22; First posted 2025-07-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gout
Keywords: Dotinurad; Allopurinol; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Allopurinol; dotinurad

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Allopurinol (Active Comparator): Participants will discontinue their allopurinol and start on study-supplied allopurinol at the same dose once a day (QD) through Week 64.
  Interventions: Drug: Allopurinol
- Dotinurad 2 mg Maintenance (Experimental): Participants will discontinue their allopurinol and start dotinurad 1 mg QD for first 4 weeks (Weeks 1-4) and then dotinurad 2 mg QD through Week 64.
  Interventions: Drug: Dotinurad
- Dotinurad 4 mg Maintenance (Experimental): Participants will discontinue their allopurinol and start dotinurad 1 mg QD for first 4 weeks (Weeks 1-4), dotinurad 2 mg QD for the next 8 weeks (Weeks 5-12), and dotinurad 4 mg QD thereafter through Week 64.
  Interventions: Drug: Dotinurad

INTERVENTIONS:
Drug: Allopurinol — Over-encapsulated tablets containing active drug substance administered orally (PO).
  Arms: Allopurinol
Drug: Dotinurad — Over-encapsulated tablets containing active drug substance administered PO.
  Arms: Dotinurad 2 mg Maintenance; Dotinurad 4 mg Maintenance

SUMMARY:
The primary objective of this study is to evaluate the efficacy of dotinurad in lowering serum uric acid (sUA) at Week 24 compared with allopurinol in adult participants with hyperuricemia associated with gout.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years of age (inclusive) at the time of signing informed consent.
2. Diagnosis of gout based on 2015 American College of Rheumatology (ACR)-European Union League Against Rheumatism (EULAR) criteria for at least 1 year.
3. Had at least 2 gout flares in the 12 months prior to Screening (reported by the participant or documented in the participant's medical records).
4. Participant must be on a stable background allopurinol dose of ≥300 mg/day (200 mg/day for those with moderate renal impairment) up to 600 mg/day for at least 3 months prior to Screening and remain on their dosing regimen until Day 1.
5. sUA level ≥6.5 mg/dL at Screening Visit 1 (Day -35 Visit) and Screening Visit 2 (Day -7 Visit).
6. Female participants of childbearing potential must have a negative serum pregnancy test at Screening Visit 1 (Day -35 Visit) and Screening Visit 2 (Day -7 Visit), a negative urine pregnancy test on Day 1, and must not be breastfeeding.
7. Fertile male participants and female participants of childbearing potential must be willing to completely abstain from heterosexual sex or agree to use acceptable contraception from the time of signing informed consent through 30 days after the last dose of study drug.

Exclusion Criteria:

1. History of or presence of kidney stones within 1 year prior to Screening.
2. History of or presence of malignancy in the last 5 years other than treated cutaneous basal or squamous cell carcinoma.
3. Hypersensitivity or intolerance to dotinurad or to colchicine and nonsteroidal anti-inflammatory drugs.
4. Known or suspected history of drug abuse, a positive drug test at Screening Visit 1, or a recent history of alcohol abuse.
5. Known history of or positive results for human immunodeficiency virus, Hepatitis B Surface Antigen, or Hepatitis C antibodies during Screening.
6. Current or historical evidence of any clinically significant disease or condition that, in the opinion of the Investigator, may compromise participant safety or study compliance or may confound interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-11-29 (Estimated); Study Completion 2027-11-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With an sUA Level <6.0 mg/dL at Week 24 | Week 24

SECONDARY OUTCOMES:
Percentage of Participants With an sUA Level <6.0 mg/dL at Weeks 16, 20 and 24 Inclusive | Weeks 16, 20 and 24
Mean Rate of Gout Flares Requiring Treatment From Week 36 Through Week 64 | Week 36 through Week 64
Percentage of Participants With an sUA level <5.0 mg/dL at Week 24 and no Gout Flares Requiring Treatment From Week 36 Through Week 64 | Week 24 and Week 36 through Week 64
Mean Change From Baseline in sUA at Week 24 | Baseline and Week 24
Percentage of Participants who do not Have a Gout Flare Requiring Treatment From Week 24 Through Week 64 | Week 24 through Week 64
Percentage of Participants With an sUA Level <6.0 mg/dL at Each Visit | Up to Week 68
Percentage of Participants With an sUA Level <5.0 mg/dL at Each Visit | Up to Week 68
Percentage of Participants With an sUA Level <4.0 mg/dL at Each Visit | Up to Week 68
Absolute Change from Baseline in sUA Levels at Each Visit | Baseline to Week 68
Percent Change from Baseline in sUA Levels at Each Visit | Baseline to Week 68
Percentage of Participants With a Gout Flare Requiring Treatment at Each Month Between Week 24 and the end of Study | Week 24 to Week 68
Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) | Day 1 through Week 68
Percentage of Participants With Serious Adverse Events (SAEs) | Day 1 through Week 68

CONTACTS AND LOCATIONS:
Locations (95):
- United States (76):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Associates (AARA) - Gilbert, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Associates (AARA) - Glendale, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Associates (AARA) - Mesa, Mesa, Arizona
  - Del Sol Research Management - Tucson East, Tucson, Arizona
  - Del Sol Research Management - Tucson, Tucson, Arizona
  - Medvin Clinical Research - Covina, Covina, California
  - West Coast Research, Dublin, California
  - Infinity Clinical Research, Norco, California
  - Amicis Research Center - Balboa, Northridge, California
  - Dream Team Clinical Research, Pomona, California
  - Velocity Clinical Research - San Bernardino, San Bernardino, California
  - Acclaim Clinical Research, Inc., San Diego, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - BTC Network - Encompass Clinical Research, Spring Valley, California
  - Cohen Medical Centers, Thousand Oaks, California
  - Medvin Clinical Research - Tujunga, Tujunga, California
  - Denver Arthritis Clinic - Lowry, Denver, Colorado
  - Bradenton Research Center, Bradenton, Florida
  - Herco Medical and Research Center, Inc, Coral Gables, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Best Quality Research, Hialeah, Florida
  - Health Awareness Inc, Jupiter, Florida
  - Clinical Research of Center Florida, Lakeland, Florida
  - Anchor Medical Research, LLC, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Omega Research DeBary, Orlando, Florida
  - D&H Pompano Research Center, Pompano Beach, Florida
  - Clinical Research Trials of Florida, Tampa, Florida
  - DelRicht Research - Atlanta, Atlanta, Georgia
  - Chicago Clinical Research Institute, Inc. (CCRII), Chicago, Illinois
  - Flourish Chicago - Ravenswood (Great Lakes Clinical Trials), Chicago, Illinois
  - Healthcare Research Network - Tinley Park, Flossmoor, Illinois
  - Investigators Research Group, Brownsburg, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Delricht Research - Better Life Direct Primary Care, Indianapolis, Indiana
  - Delricht Research - Concierge And Direct Primary Care, Overland Park, Kansas
  - DelRicht Research - Louisville (Derby City DPC), Louisville, Kentucky
  - Tandem Clinical Research - Metairie Clinic, Metairie, Louisiana
  - DelRicht Research - LCMC Health Urgent Care - Lakeview, New Orleans, Louisiana
  - DelRicht Research - Prairieville, Prairieville, Louisiana
  - MD Medical Research - Oxon Hill, Oxon Hill, Maryland
  - DelRicht Research - Maryland (Matthew L. Mintz, MD, FACP), Rockville, Maryland
  - MedVadis Research, Waltham, Massachusetts
  - Clinical Research Institute of Michigan - St. Clair Shores, Saint Clair Shores, Michigan
  - DM Clinical Research - Detroit, Southfield, Michigan
  - Oakland Medical Center, Troy, Michigan
  - Healthcare Research Network, Hazelwood, Missouri
  - Delricht Research - Command Family Medicine, Springfield, Missouri
  - DelRicht Research - Town and Country, Town and Country, Missouri
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Ellipsis Research Group, Brooklyn, New York
  - New York University Langone Orthopedic Center, New York, New York
  - DelRicht Research - Charlotte (Direct Primary Care - DPC), Charlotte, North Carolina
  - Carteret Medical Group LLC, Morehead City, North Carolina
  - Shelby Clinical Research, LLC - North Carolina, Shelby, North Carolina
  - Hometown Urgent Care and Research - Dayton, Dayton, Ohio
  - Delricht Research - Concierge Medicine Of Cincinnati, Mason, Ohio
  - DelRicht Research - Tulsa, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Suburban Research Associates - West Chester Office, West Chester, Pennsylvania
  - Coastal Carolina Research Center - Main, North Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - DelRicht Research - Hendersonville, Hendersonville, Tennessee
  - Zenos Clinical Research, Dallas, Texas
  - Lone Star Arthritis & Rheumatology Associates - Denton, Denton, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Alliance Clinical Lewisville (Epic Clinical Research), Lewisville, Texas
  - Southwest Rheumatology Research, Mesquite, Texas
  - Discovery Clinical Trials, San Antonio, Texas
  - ERG - Endeavor Clinical Trials, San Antonio, Texas
  - DM Clinical Research - Tomball - Multiple Specialties, Tomball, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
- Poland (12):
  - Centrum Medyczne Solumed, Poznan, Greater Poland Voivodeship
  - FutureMeds - Krakow, Krakow, Lesser Poland Voivodeship
  - FutureMeds - Wroclaw, Wroclaw, Lower Silesian Voivodeship
  - Innova Clinic, Plońsk, Masovian Voivodeship
  - Prolato Clinical Research Center, Sochaczew, Masovian Voivodeship
  - Medicover Integrated Clinical Services- MICS Centrum Medyczne Warszawa Chlodna, Warsaw, Masovian Voivodeship
  - FutureMeds - Targówek, Warsaw, Masovian Voivodeship
  - ClinicMed Daniluk, Nowak Spółka Komandytowa, Bialystok, Podlaskie Voivodeship
  - FutureMeds Gdynia, Gdynia, Pomeranian Voivodeship
  - Med-Progress Ośrodek Nowoczesnego Leczenia, Wejherowo, Pomeranian Voivodeship
  - Pro Familia - Katowice, Katowice, Silesian Voivodeship
  - Silmedic sp. z o.o., Katowice, Silesian Voivodeship
- Spain (7):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Clínica Gaias Santiago, Santiago de Compostela, La Coruña
  - Accellacare - Alcobendas, Alcobendas, Madrid
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
  - Hospital Quirónsalud Infanta Luisa, Seville, Sevilla
  - Clínica NTDE - Nuevas Tecnologías en Diabetes y Endocrinología, Seville, Sevilla
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported for publication, after deidentification.
Supporting Information: Study Protocol, SAP